CLINICAL TRIAL: NCT00682825
Title: BAG-RECALL Study: BIS or Anesthesia Gas to Reduce Explicit Recall
Brief Title: Study Evaluating Whether the Bispectral Index Prevents Patients at Higher Risk From Being Awake During Surgery and Anesthesia
Acronym: BAG-RECALL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other); American Society of Anesthesiologists (Other); University of Chicago (Other); University of Manitoba (Other); University of Michigan (Other)
Responsible Party: Michael Avidan, Washington University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-1253
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Explicit Recall of Intra-Operative Events
Keywords: Anesthesia; Awareness; Bispectral; BIS; Recall

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Bispectral index-guided protocol
  Interventions: Behavioral: Bispectral index protocol
- 2 (Active Comparator): End-tidal anesthetic gas-guided protocol
  Interventions: Behavioral: End tidal anesthetic gas-guided

INTERVENTIONS:
Behavioral: Bispectral index protocol — Aim to titrate anesthesia to maintain BIS between 40 and 60.
  Arms: 1
Behavioral: End tidal anesthetic gas-guided — Aim to maintain anesthetic gas between 0.7 and 1.3 MAC equivalents
  Arms: 2

SUMMARY:
The overall purpose of this study is to see if a Bispectral Index (BIS) monitor, a Food and Drug Administration (FDA) approved brain monitoring device, will help to reduce the risk of patients remembering being awake during surgery. The BIS monitor may be able to measure how asleep a patient is during surgery. Using the BIS monitor to guide anesthesia will be compared with using the concentration of anesthetic gas to guide anesthesia.

DETAILED DESCRIPTION:
The incidence of anesthesia awareness (AA) is 0.1-0.2% and may result in post traumatic stress disorders. For some patients, owing to illness, medications, substance misuse or surgery, the risk approaches 1%. The B-AWARE Study by Myles et al. suggested that the bispectral index (BIS) monitor, which reportedly reflects anesthetic depth, may decrease the incidence of AA in higher risk patients by 82%. The American Society of Anesthesiologists has published a practice advisory on AA, which does not recommend the routine use of cerebral function monitors. We propose to test the hypothesis that an anesthetic protocol based on BIS decreases the incidence of AA among higher risk patients compared with an anesthetic protocol based on the end-tidal anesthetic gas (ETAG) concentration. We have completed a randomized, single-blinded prospective feasibility study (The B-Unaware Trial) which enrolled 2000 patients at higher risk for AA. Four patients (0.21%; 95% CI=0.06% to 0.57%) had definite AA, of whom two were in the BIS-guided group and two in the ETAG-guided group. Nine patients (0.46%; 95% CI=0.22% to 0.91%) had definite or possible AA, of whom six were in the BIS-guided group and three in the ETAG-guided group. The BAG RECALL study will be a multi-center, prospective, single-blinded, randomized study enrolling 6000 patients at higher risk for AA. The BAG RECALL study is adequately powered and rigorously designed to answer with a reasonable degree of scientific probability whether BIS guidance results in clinically relevant reduction in anesthesia awareness among higher risk patients undergoing general anesthesia.

At the University of Michigan, a parallel study will be conducted - Michigan Awareness Control Study, MACS (NCT00689091) - enrolling 30,000 patients to assess whether the BIS monitor decreases the likelihood of anesthesia awareness among all patients undergoing general anesthesia, regardless of their risk profile. The investigators of this study and the BAG-RECALL study have collaborated in designing these studies and are pre-specifying that common outcome measures will be examined collaboratively including data from both studies.

ELIGIBILITY:
Inclusion Criteria:

MUST HAVE:

General Anesthesia with volatile anesthetic

PATIENT CHARACTERISTICS

Major Criteria (Must have any 1 of the following:)

1. Planned open heart surgery
2. Medications - anticonvulsants, abuse of opiates, benzodiazepines, cocaine
3. EF<40%
4. Prior history of awareness (recall)
5. History of difficult intubation or anticipated difficult intubation
6. ASA IV or V status
7. Aortic stenosis
8. End stage lung disease
9. Marginal exercise tolerance not secondary to musculoskeletal dysfunction
10. Pulmonary hypertension
11. Daily alcohol consumption

Exclusion Criteria:

1. Surgical procedure that prevents the use of the BIS (e.g. surgery of forehead)
2. Patient positioning prevents use of the BIS
3. Surgery with wake-up test.
4. Less than 18 years of age
5. Vulnerable populations, such as those with dementia and those unable to provide informed consent.
6. Stroke with residual neurological deficits

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The incidence of explicit recall of events during the surgical and anesthetic periods. | Three years

SECONDARY OUTCOMES:
Meta-analysis for anesthesia awareness incorporating higher risk patients from the completed B-Unaware Trial (NCT00281489), the BAG-RECALL Trial, and the Michigan Awareness Control Study (MACS)(NCT00689091). | Three years
Incidence of post-traumatic stress disorder (PTSD). | Five years
Association between type of awareness event and PTSD, and whether the PTSD is associated with late reporting (30 days) of awareness. | 5 years
Types of dreams and their relationship to BIS and ETAG. | Three years
The relationship between deep hypnotic time, anesthetic dose (MAC), mean arterial pressure, and end tidal carbon dioxide, and early (one-month) and late (one-year) mortality. | Four years
Relationship between BIS, heart rate and blood pressure. | Three years
Relationship between BIS and anesthesia dose and concentration. | Three years
Association between baseline BIS values, patient health and early (one-month) and late (one-year) mortality. | Four years
Interaction between hemispheric dominance and BIS. | Three years
Effect of red hair phenotypes on the relationship between ETAG and BIS. | Three years
Refinement of risk factors for anesthesia awareness. | Three years
Relationship between rising BIS in the PACU and first memory after surgery. | Three years
Postoperative delirium. | Three years
BIS and mixed venous saturation. | Three years
Induction of anesthesia and hypotension. | Three years
Incidence of postoperative nausea and vomiting. | Three years
Incidence of and severity of postoperative pain. | Three years
Effect of BIS and ETAG protocols on time to open eyes, time to extubation, and time spent in the postoperative recovery unit. | Three years
Effect of a defasciculating dose of a non-depolarizing muscle relaxant on BIS. | Three years
The effect of patient temperature on BIS. | Three years
Incidence of recall of traveling to the OR among patients who receive midazolam in the holding area and whose initial BIS reading in the OR is > 60. | Three years
Relationship between BIS, ETAG and EEG parameters. | Three years
Annual assessment of practitioners' abilities to interpret BIS tracings and to identify artefacts. | Three years
Differences in anesthesia practice among four institutions in the USA and Canada as judged by anesthetic doses and BIS readings. | Three years
Effect of BIS and ETAG protocols on anesthetic dose administration and on BIS readings. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBCh FCA, Principal Investigator — Washington University School of Medicine; David Glick, MD, Study Director — University of Chicago; Eric Jacobsohn, MBChB, Study Chair — University of Manitoba; Michael O'Connor, MD, Study Director — University of Chicago; Alex S Evers, MD, Study Chair — Washington University School of Medicine
Locations (3):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Washington University, St Louis, Missouri
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Avidan MS, Palanca BJ, Glick D, Jacobsohn E, Villafranca A, O'Connor M, Mashour GA; BAG-RECALL Study Group. Protocol for the BAG-RECALL clinical trial: a prospective, multi-center, randomized, controlled trial to determine whether a bispectral index-guided protocol is superior to an anesthesia gas-guided protocol in reducing intraoperative awareness with explicit recall in high risk surgical patients. BMC Anesthesiol. 2009 Nov 30;9:8. doi: 10.1186/1471-2253-9-8. PMID 19948045
- [Background] Mashour GA, Tremper KK, Avidan MS. Protocol for the "Michigan Awareness Control Study": A prospective, randomized, controlled trial comparing electronic alerts based on bispectral index monitoring or minimum alveolar concentration for the prevention of intraoperative awareness. BMC Anesthesiol. 2009 Nov 5;9:7. doi: 10.1186/1471-2253-9-7. PMID 19891771
- [Background] Mashour GA, Esaki RK, Tremper KK, Glick DB, O'Connor M, Avidan MS. A novel classification instrument for intraoperative awareness events. Anesth Analg. 2010 Mar 1;110(3):813-5. doi: 10.1213/ANE.0b013e3181b6267d. Epub 2009 Aug 27. PMID 19713251
- [Derived] Willingham M, Ben Abdallah A, Gradwohl S, Helsten D, Lin N, Villafranca A, Jacobsohn E, Avidan M, Kaiser H. Association between intraoperative electroencephalographic suppression and postoperative mortality. Br J Anaesth. 2014 Dec;113(6):1001-8. doi: 10.1093/bja/aeu105. Epub 2014 May 22. PMID 24852500
- [Derived] Whitlock EL, Torres BA, Lin N, Helsten DL, Nadelson MR, Mashour GA, Avidan MS. Postoperative delirium in a substudy of cardiothoracic surgical patients in the BAG-RECALL clinical trial. Anesth Analg. 2014 Apr;118(4):809-17. doi: 10.1213/ANE.0000000000000028. PMID 24413548
- [Derived] Avidan MS, Jacobsohn E, Glick D, Burnside BA, Zhang L, Villafranca A, Karl L, Kamal S, Torres B, O'Connor M, Evers AS, Gradwohl S, Lin N, Palanca BJ, Mashour GA; BAG-RECALL Research Group. Prevention of intraoperative awareness in a high-risk surgical population. N Engl J Med. 2011 Aug 18;365(7):591-600. doi: 10.1056/NEJMoa1100403. PMID 21848460
- See also: Bispectral Index (BIS) Versus Electronic Alerts in the Prevention of Awareness (MACS) — http://www.clinicaltrials.gov/ct2/show/NCT00689091